CLINICAL TRIAL: NCT04706299
Title: Effects of Surgical Mask Use on Peak Torque, Total Work and Interset Fatigability During Isokinetic Strength Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Matthew Kampert, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20-1303
Record Dates: First submitted 2021-01-10; First posted 2021-01-12 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Prevention of COVID-19
Keywords: Exercise; Face Mask; COVID-19; Resistance Training
MeSH Terms: conditions — Motor Activity; COVID-19 | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This is a prospective study conducted using a randomized-control crossover design where participants will complete resistance exercise (RE) protocol utilizing a Biodex System 4 and Advantage V5 software with a standard leg attachment, on 2 separate days with at least 48 hours and no greater than seven days between tests.
Masking Description: Participants will perform a RE protocol under 2 different conditions, once without a mask and once while wearing a surgical mask. A coin flip wil be utlize to minimize the possibility of familiarization or training effects, and maintain complete randomness of the assignment of which RE conditions is performed first, in addition to which leg is tested first. This simple randomization method to determine the assignment will follow (heads = No mask, tails = surgical mask and heads = dominant leg 1st, tails = nondominant leg 1st, on the 1st and 2nd coin toss, respectively). Study participants will be asked which leg they prefer to kick a ball with to identify their dominant leg for data collection purposes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Mask (Active Comparator): Will not wear a mask
  Interventions: Other: Resistance Exercise
- Surgical mask (Experimental): Will wear a surgical nose and face covering
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Other: Resistance Exercise — Participants will perform for each leg, 3 sets comprised of 15 repetitions set to 180 degrees per second of an isokinetic, concentric knee extension and flexion. Resulting in a 20 second long working set (10 seconds extension, 10 seconds flexion), per set. Each set will be followed by a 90 second period of recovery. After completing 3 sets on initial leg, testing will be set up for second leg.

SUMMARY:
The coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is highly transmittable person-to-person when an infected individual coughs, sneezes or talks while within at least 6 feet (1.8 m) of a neighboring individual. Guidelines set forth by the Centers for Disease Control and Prevention (CDC) state that nose and mouth facial coverings are recommended at all levels for source control as a simple barrier to help prevent respiratory droplet transmission. It is important to remember that increased viral shedding occurs during elevated ventilatory rates that are observed during exercise within a shared space, such as gyms or fitness studios increase the rate of transmission. However, there is limited research studying the effects of mask use during exercise, and no research evaluating these effects specifically during resistance-based exercise. Therefore, the purpose of this investigation is to examine the effects of wearing a surgical face mask while performing resistance exercise on average peak force, total work, heart rate (HR), oxygen saturation (SpO2) and breathing discomfort.

DETAILED DESCRIPTION:
Despite the accumulating evidence supporting the favorable impact and potentially life-saving benefits of routine public mask wearing has on lowering the risk of COVID-19 transmission, recommendations for mask use have been met with resistance by some individuals. With the numerous health benefits greatly outweighing the document complaints of discomfort and headaches, it becomes puzzling why there is not universal support for these recommendations made by experts. Additional insight to this ongoing issue is provided in an extremely informative commentary provided by Scheid et al, in which they present theoretical evidence suggesting that there may be consequential psychological impacts of mask wearing on the basic psychological needs of competence, autonomy, and relatedness. Which may contribute to the controversy associated with mask use. It is also important to consider that such subjective experiences caused by mask wearing have been demonstrated to be exacerbated when physical exertion is performed at intensities above activities of daily living, such as during incremental aerobic or resistance exercise.

Currently, the CDC identifies age > 65, BMI > 30, diabetes, smoking, chronic obstructive pulmonary disease, heart conditions, or an immunocompromised state as risk factors for severe illness from COVID-19. Research conducted by Barkley et al, revealed that university closure increased sedentary behavior in all study participants, but only decreased physical activity in individuals who were the most active pre-cancellation. Highlighting concerns that pandemic-related closure of facilities such as gyms, which are designed for physical activity may disproportionately impact a more active population. Increased sedentary behavior and reduced physical activity will likely exacerbate these known risk factors for severe illness from COVID-19, and contribute to overloading our healthcare systems . While it is still recommended that adults of all ages should achieve 150-300 minutes of moderate or 75-150 minutes of vigorous (or an equivalent combination) physical activity per week, along with at least 2 days per week of muscle strengthening activities. Unfortunately, evidence based guidelines have not yet been developed to guide universal mask use during exercise and sporting events.

In this proposed randomized controlled cross-over study, we aim to evaluate in non-COVID-19 infected and otherwise healthy young-to-middle aged adults whether compared with performing resistance exercise (RE) with no mask (NM), 1) are there effects of wearing a surgical mask on physiological or psychological responses during RE that limit peak force or work performed in an exercise session, and 2) does wearing a surgical mask during resistance exercise yield clinically relevant and dangerous absolute indications warranting early exercise termination. Isokinetic testing can be used to provide valid, reliable, objective measure of a muscle's performance and offers significant clinical controls to simulate a resistance training workout. The lever arm speed measuring muscular output by the participant can be adjusted depending on the desired number of repetitions or duration test performed. Various skeletal muscle metabolic systems could be stressed depending on the effort and duration of time under tension, making it an efficient and reliable method for the assessment of muscle performance under various environmental conditions, including wearing a mask during a resistance training workout. To our knowledge this is the first study to assess the effects of wearing protective nose and face covering on resistance exercise capacity, estimate arterial oxyhemoglobin saturation (SpO2), and degree of discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Study inclusion criteria required potential participants must be apparently healthy without a history of any chronic disease (including absence of exercise induced asthma),
* Asymptomatic and without previous positive COVID-19 test
* Demonstrate no orthopedic or medical limitation that could be the cause of exercise termination

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of wearing a surgical face mask while performing resistance exercise on average peak force and total work performed. | 1 week
  For this we will utilize the Biodex system to measure average peak torque (highest force output in a repetition) and total work (muscle's cumulative ability to produce force throughout range of motion for the entire set of repetitions). Working Hypothesis: There will not be a statistically significant difference of peak torque and total work while wearing a mask compared without a mask.

SECONDARY OUTCOMES:
Identify changes in the level of discomfort experienced while wearing a surgical mask during resistance exercise. | 1 week
  For this, subjective experience of wearing or not wearing a facial covering will be evaluated at both pre and post- exercise utilizing a perceptions instrument questionnaire (12,16,20). Working hypothesis: Participants performing resistance training while wearing surgical mask covering their nose and mouth with experience an increased perception of elevated breathing resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kampert, Principal Investigator — Staff Physician
Locations (1):
- Cleveland Clinic Sports Health, Garfield Heights, Ohio, United States

IPD SHARING:
Plan to Share IPD: No